CLINICAL TRIAL: NCT04135209
Title: Evaluation of Macular Microvasculature in High Myopia Using Optical Coherence Tomography Angiography
Brief Title: Optical Coherence Tomography Angiography in Myopic Patients
Status: Completed | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, M. Tarek A. Moustafa, Lecturer of Ophthalmology, Minia University
Other Study IDs: 68-7/2018
Record Dates: First submitted 2019-10-12; First posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Myopia
Keywords: Optical coherence tomography; Angiography; Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy controls: Healthy individuals of age-matched
  Interventions: Diagnostic Test: Optical coherence tomography angiography OCTA
- Myopic patients: Patients with myopia who meet the inclusion criteria
  Interventions: Diagnostic Test: Optical coherence tomography angiography OCTA

INTERVENTIONS:
Diagnostic Test: Optical coherence tomography angiography OCTA — Macular scanning using regular structural OCT as well as microvasculature analysis using OCTA
  Other Names: OCTA

SUMMARY:
The aim of this study is to investigate the macular microvascular network alterations in high myopic eyes using optical coherence tomography angiography.

DETAILED DESCRIPTION:
High myopia is defined as a refractive error equal to or more than -6 D, and/or axial length equal to or more than 25.5 mm².Axial elongation of the globe and subsequent stretch of the retina leads to sight threatening complications.

Quantitative measurements of retinal vasculature in the healthy eye have been reported using several in vivo and in vitro techniques, including confocal microscopy, fluorescein angiography (FA), and swept-source optical coherence tomography (ssOCT) angiography.

The aim of this study is to investigate the macular microvascular network alterations in high myopic eyes using optical coherence tomography angiography.

This cross-sectional prospective study included 75 eyes of 54 patients, they were recruited from the outpatient clinic of ophthalmology department of El-Minia university hospital.They were divided into two groups, group A included 25 normal eyes of 25 patients. Group B included 50 myopic eyes of 30 patients.

All patients subjected to history taking and full ophthalmological examination in addition to axial length measurment before performing OCTA.

ELIGIBILITY:
Inclusion Criteria:

* • Highly myopic subjects, defined as those with spherical equivalents (SEs) of -6 or more, with axial length greater than 26.5 mm.

Group B individuals were chosen among healthy age-matched controls.

Exclusion Criteria:

* • Patients younger than 18 years old, or older than 45 years.

  * Any patient with macular pathology (e.g. diabetic retinopathy, hypertensive retinopathy, dystrophy)
  * Myopic patients with any vitro-retinal abnormalities (e.g. choroidal neovascular membrane (CNVM), foveoschisis,macular hole)
  * Patients who underwent previous intra ocular surgical procedures.
  * Patients with previous history of intraocular injections.
  * Glaucomatous patients.

Exclusion criteria to the images that has been captured:

* - Low signal strength index (less than 50).
* - Presence of blink artefacts.
* - Poor fixation leading to motion or doubling artefacts.
* - Media opacity obscuring view of the vasculature.
* - Segmentation error due to cystoid macular oedema or epi-retinal membrane, among others.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Groiup A patients were chosen when met the inclusion criteria. Group B individuals were chosen among healthy age-matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Difference in angiography between the 2 groups | through study completion, an average of 4 weeks
  The difference of the volumetric data generated automatically from the OCTA machine at the 3 levels, (the inner retina, outer retina and the choriocapillaris) in three zones (the fovea, the parafovea and the whole image)

CONTACTS AND LOCATIONS:
Overall Officials: M. Tarek A Mosutafa, MD, Principal Investigator — Lecturer of ophthalmology
Locations (1):
- Minia University, Minya, Minya Governorate, Egypt